CLINICAL TRIAL: NCT05018195
Title: Profile of Adipocytokines in Patients With Endometrial Cancer: Focus on Various Types of Adipose Tissues
Brief Title: Adipocytokines in Endometrial Cancer
Acronym: ACEmCa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202106074RIND
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Endometrial Cancer
Keywords: Obesity; Inflammation; Adiponectin; Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms; Obesity; Inflammation

STUDY DESIGN:
Intervention Model Description: Two groups: women receive surgery for benign gynecologic lesions and women receive surgery for endometrial cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benign (Active Comparator): Women who receive surgery for benign lesions including leiomyoma, adenomyosis, or ovarian cysts. We will obtain one 5*5 cm omental fat and one 3*3 cm subcutaneous adipose tissue during surgery.
  Interventions: Procedure: Excise adipose tissue
- Endometrial cancer (Experimental): Women who receive surgery(staging or cytoreductive surgery) for endometrial cancer. We will obtain one 5*5 cm omental fat and one 3*3 cm subcutaneous adipose tissue during surgery.
  Interventions: Procedure: Excise adipose tissue

INTERVENTIONS:
Procedure: Excise adipose tissue — Perform partial omentectomy to obtain one 5*5 cm omental fat and excise one 3*3 cm subcutaneous adipose tissue( 2 finger width above the pubic symphysis) during surgery

SUMMARY:
Endometrial cancer incidence rates were increasing in the past two decades with a continuous rising trend in Taiwan. Uterine cancer was attributable to obesity based on their association with excess body weight in most epidemiological cohort studies. However, the prevalence of obesity was lower in Taiwan.Therefore, we will study if adipose tissues depots in different locations of body could reflect or correlate the pathogenesis of endometrial cancer.

DETAILED DESCRIPTION:
Besides lipid metabolism, adipose tissue plays import roles in regulation of hormones, adipokines, cytokines and immunocytes. Adipose tissue is now known as endocrine organ which to express and secrete a variety of bioactive peptides, known as adipokines. We will evaluate the difference various adipocytokines between visceral and subcutaneous adipose tissues between women with benign lesions and endometrial cancer. We will study the inter-individual differences in adipocytokines between two types of adipose tissues and their correlation with image quantification.

ELIGIBILITY:
Inclusion Criteria:

Women diagnosed with primary endometrial cancer and undergo surgery, with or without adjuvant therapy in our hospital (EmCa group); women received surgery for benign pelvic lesions in our hospital (control group)

Exclusion Criteria:

Women with an underlying malignancy or any concomitant malignancy, prior chemotherapy or radiation before diagnosis of endometrial cancer, history of autoimmune diseases or immunosuppressive agent use

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women received gynecologic surgery
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-07-29 (Estimated); Study Completion 2022-07-29 (Estimated)

PRIMARY OUTCOMES:
Adipocytokines profile | During operation
  Adipocytokines including leptin, adiponectin, visfatin, resistin, omentin, IL-1β, IL-6, IL-8, IL-10, TNF-α, IFNγ

IPD SHARING:
Plan to Share IPD: Undecided
Share the adipocytokines profile raw data

REFERENCES:
- [Result] Sung H, Siegel RL, Torre LA, Pearson-Stuttard J, Islami F, Fedewa SA, Goding Sauer A, Shuval K, Gapstur SM, Jacobs EJ, Giovannucci EL, Jemal A. Global patterns in excess body weight and the associated cancer burden. CA Cancer J Clin. 2019 Mar;69(2):88-112. doi: 10.3322/caac.21499. Epub 2018 Dec 12. PMID 30548482
- [Result] Lin YC, Yen LL, Chen SY, Kao MD, Tzeng MS, Huang PC, Pan WH. Prevalence of overweight and obesity and its associated factors: findings from National Nutrition and Health Survey in Taiwan, 1993-1996. Prev Med. 2003 Sep;37(3):233-41. doi: 10.1016/s0091-7435(03)00119-1. PMID 12914829
- [Result] Chen LJ, Fox KR, Haase A, Wang JM. Obesity, fitness and health in Taiwanese children and adolescents. Eur J Clin Nutr. 2006 Dec;60(12):1367-75. doi: 10.1038/sj.ejcn.1602466. Epub 2006 Jun 14. PMID 16775581
- [Result] Lai JC, Weng CS, Huang SM, Huang N, Chou YJ, Wang CC, Wang KL. Incidence and lifetime risk of uterine corpus cancer in Taiwanese women from 1991 to 2010. Taiwan J Obstet Gynecol. 2017 Feb;56(1):68-72. doi: 10.1016/j.tjog.2015.09.010. PMID 28254229
- [Result] Hopkins BD, Goncalves MD, Cantley LC. Obesity and Cancer Mechanisms: Cancer Metabolism. J Clin Oncol. 2016 Dec 10;34(35):4277-4283. doi: 10.1200/JCO.2016.67.9712. Epub 2016 Nov 7. PMID 27903152
- [Result] Rakotoarivelo V, Lacraz G, Mayhue M, Brown C, Rottembourg D, Fradette J, Ilangumaran S, Menendez A, Langlois MF, Ramanathan S. Corrigendum to "Inflammatory cytokine profiles in visceral and subcutaneous adipose tissues of obese patients undergoing bariatric surgery reveal lack of correlation with obesity or diabetes" EBioMedicine 30C (2018) 237-247. EBioMedicine. 2018 Nov;37:564-568. doi: 10.1016/j.ebiom.2018.10.025. Epub 2018 Oct 16. No abstract available. PMID 30341040